CLINICAL TRIAL: NCT05229237
Title: A Multicenter, Observational, Registrie Study of Conbercept in the Treatment of Polypoidal Choroidal Vasculopathy（START Study）
Brief Title: Conbercept for Polypoidal Choroidal Vasculopathy（START Study）
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: START
Record Dates: First submitted 2018-04-18; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2018-04

CONDITIONS: Polypoidal Choroidal Vasculopathy; Conbercept
Keywords: registration study; Polypoidal Choroidal Vasculopathy; Conbercept
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy | interventions — KH902 fusion protein

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Conbercept — Intravitral injection of Conbercept (0.5 mg/0.05 mL, Chengdu Kanghong Biotech, Inc.)
  Other Names: This was no other intervention name

SUMMARY:
1. To evaluate the effectiveness of Conbercept for PCV patients.
2. To describe the characteristics of PCV.
3. To describe the adverse events (AE) of Conbercept in the treatment of PCV.
4. Todescirbe the real situation and prognosis of PCV patients in our country.

DETAILED DESCRIPTION:
1. To observe the visual changes in PCV patients receiving Conbercept treatment, so as to evaluate the effectiveness of the treatment. Changes of OCT, ICGA, quality of life and visual function would be observed and evaluated.
2. To observe and describe the characteristics of PCV.
3. To observe and describe the incidence of adverse events (AE) and serious adverse events (SAE) of Conbercept in the treatment of PCV, so as to evaluate the safety of this treatment.
4. To observe and descirbe the real situation and prognosis of PCV patients in our country.

ELIGIBILITY:
Inclusion Criteria:

* According to the current diagnostic criteria, diagnosed as PCV patients
* Conbercept is used for treatment, and the recommended treatment scheme is 3+PRN
* Local and systemic anti-VEGF therapy was not used for at least three months before enrollment
* The patient volunteers to take part in this observational study, and signs the informed consent
* The patient can follow-up regularly (at least 4 times of follow-up in one year)

Exclusion Criteria:

* The patient has serious systemic disease, and the current clinical treatment is contraindicated
* Local or systemic anti-VEGF therapy was used for less than three months before enrollment
* Existence of diseases unsuitable to accept intravitreal Conbercept, including uncontrolled hypertension and diabetes, AIDS, malignant tumors, active hepatitis, severe renal failure, severe mental, nerve, cardiovascular, respiratory and immune diseases
* During six months before screening, there were cardiovascular events such as stroke, transient ischemic attack, myocardial infarction or acute congestive heart failure
* Ocular contraindications, including active intraocular inflammation, infectious endophthalmitis, corneal ulcer, scleritis, uncontrolled glaucoma and so on
* Patients who could not follow up regularly
* Patients who refuse to sign the informed consent
* Others

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed as polypoid choroidal vasculopathy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-06-05 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 6 months after the first Conbercept treatment
  Best corrected visual acuity using ETDRS chart (letter numbers)

SECONDARY OUTCOMES:
OCT and OCTA | 12 months after the first Conbercept treatment
  Changes of central retinal thickness and size of PED (μm)
FFA&ICGA | 12 months after the first Conbercept treatment
  Changes of PCV lesions on ICGA (μm)

CONTACTS AND LOCATIONS:
Overall Officials: Youxin Chen, Professor, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided